CLINICAL TRIAL: NCT02724475
Title: Laser Ablation for Intermediate and Advanced Hepatocellular Carcinoma With Portal Vein Tumor Thrombus: A Randomized Controlled Trial
Brief Title: Laser Ablation for Intermediate and Advanced Hepatocellular Carcinoma With Portal Vein Tumor Thrombus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012ZX10002016003
Record Dates: First submitted 2016-03-28; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma; Laser Ablation; Portal Vein Tumor Thrombus
Keywords: Laser Ablation; Portal Vein Tumor; Thrombus
MeSH Terms: conditions — Carcinoma, Hepatocellular; Thrombosis | interventions — Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LA group (Experimental): Ultrasound-guided puncture to the front of the thrombus with a power of 30 watts and pulse time of 0.3-0.4 seconds with 1 second interval until the thrombus was totally eliminated.
  Interventions: Procedure: LA
- 3D-CRT group (Experimental): γ-knife treatment with radiation dose of 48-63 Gy/6-9 times.
  Interventions: Procedure: 3D-CRT

INTERVENTIONS:
Procedure: LA — Ultrasound-guided puncture to the front of the thrombus with a power of 30 watts and pulse time of 0.3-0.4 seconds with 1 second interval until the thrombus was totally eliminated
  Arms: LA group
Procedure: 3D-CRT — γ-knife treatment with radiation dose of 48-63 Gy/6-9 times
  Arms: 3D-CRT group

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most-common cancer worldwide and the second most-common cause of cancer mortality. Liver resection is the first-line curative treatment for huge HCC. The 5-year overall survival (OS) rates after hepatic resection were range from 25% to 45% and the incidence of portal vein tumor thrombus (PVTT) for intermediate and advanced hepatocellular carcinoma patients were as high as 60%-90%. At present, there is no effective treatment for patients with PVTT. Laser ablation (LA) showed a good performance in eliminating the PVTT and the three-dimensional conformal radiotherapy (3D-CRT) with γ Ray (γ-knife) can also be used to treat patients with PVTT. But there still lack of evidence-based research to compare the clinical outcome of 3D-CRT with γ Ray and LA. In view of this, we aim to implement a randomized controlled study to find out an effective treatment for intermediate and advanced hepatocellular carcinoma patients with PVTT based on evidence-based research.

ELIGIBILITY:
Inclusion Criteria:

1. Child-Pugh class B liver function；
2. Preoperative ECOG criteria score of 0-2;
3. Patients preoperatively diagnosed of hepatocellular carcinoma according to chest computed tomography (CT) and/or magnetic resonance imaging (MRI);
4. Tumor thrombus in the second-order or more peripheral branch of portal vein;
5. Tumor number ≤5 and the sum of largests tumor diameter ≤15 cm;
6. The expected survival time >6 months.

Exclusion Criteria:

1. Other anticancer treatment before treatment
2. Patients with apparent major organs (i.e. cardiac, pulmonary, cerebral and renal) dysfunction, which may affect the treatment of liver cancer
3. Patients with other diseases that may affect the treatment of this treatment
4. History of other malignant tumors
5. Patients who are participating in other clinical trials
6. Pregnant, lactating women

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Toxic and side effects caused by 3D-CRT or LA | 3 years
Postoperative complication | 3 years
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China